CLINICAL TRIAL: NCT04309942
Title: An Evaluation Study on the Performance of a Guided Clinical Pharmacy Consultation for Patients With Multiple Myeloma Following Their First Oral Anticancer Treatment
Brief Title: Evaluation Study on Performance of Guided Clinical Pharmacy Consultation in Patients With Multiple Myeloma on First Oral Anticancer Treatment
Acronym: CPS MYELOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Centre hospitalier de Perpignan (Other); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2018-01/MF
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Oral anticancer treatment; Observance
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Multicentric, prospective, randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Clinical Pharmacy Consultation group (Experimental): Patients following either Revlimid - Velcade - Dexamethasone or Revlimid - Dexamethasone protocols with the benefit of a Guided Clinical Pharmacy Consultation before beginning oral anticancer treatment for multiple myeloma.
  Interventions: Other: Guided Clinical Pharmacy Consultation
- Standard group (No Intervention): Patients following either Revlimid - Velcade - Dexamethazone or Revlimid - Dexamethazone protocols but without the benefit of a Guided Clinical Pharmacy Consultation before beginning oral anticancer treatment for multiple myeloma.

INTERVENTIONS:
Other: Guided Clinical Pharmacy Consultation — These patients will have the benefit of a Guided Clinical Pharmacy Consultation
  Arms: Guided Clinical Pharmacy Consultation group

SUMMARY:
Nowadays, more and more patients are receiving anticancer treatment by mouth and oral chemotherapy is a challenge for our health system as patients become autonomous and responsible for following their oral anti-cancer treatment at home.

According to the French National Cancer Institute around 5.000 new cases of multiple myeloma (MM) are detected each year, and this figure is on the increase. It is more common in people aged over 70. The patterns of oral anticancer medication for multiple myeloma are complex and these patients do not always follow their treatment correctly. A clinical pharmaceutical consultation guide was designed to overcome this problem.Our hypothesis is that the guided consultation would minimize the rate of discrepancies observed compared with the usual, standard type of management.

The main objective is therefore to evaluate the performance of this guided consultation (interventional group) in comparison with a control group (standard management) for patients with multiple myeloma on their first cure of oral anticancer medication.

DETAILED DESCRIPTION:
Nowadays, more and more patients are receiving anticancer treatment by mouth. In this context, the development of oral chemotherapy represents a challenge to our health system as it means adapting the hospital's organization and making it safer to manage patients who are becoming autonomous and responsible for following their oral anti-cancer treatment at home.

According to the French National Cancer Institute, around 5,000 new cases of multiple myeloma (MM) are detected each year, and this figure is on the increase year by year. It is more common in people aged over 70. Patients treated have several risk factors for not respecting medication adherence such as age, polypharmacy related to the presence of other chronic pathologies, and associated comorbidities. Furthermore, the patterns of administering oral anticancer medication for multiple myeloma are complex.

In a previous study we designed a clinical pharmaceutical consultation guide with a view to improving patients' adherence to their oral anticancer treatment. This guide was designed and validated by a multidisciplinary workgroup to ensure that it was readable, understandable and easy to memorize for the patients being treated for multiple myeloma. The guide was designed so that the information given was reproducible from one patient to another, whoever the pharmacist might be, by standardizing the information given. Our hypothesis is that the guided consultation would make it possible to minimize the rate of discordance observed compared with the usual, standard type of management.

The main objective of this study is to evaluate the performance of the guided consultation (Intervention) by evaluating the rate of discrepancies observed compared with the theoretical therapeutic pattern prescribed, compared with a control group(standard management) for patients with multiple myeloma on their first cure of oral anticancer medication.

Secondary objectives are:

A. For both groups in the study, evaluate the patients' level of knowledge and understanding of their treatment.

B. In the interventional group, evaluate the acceptability of the intervention by the patient.

C. For both groups in the study, evaluate the attitude of the patients when faced with intercurrent events (foreseeable with oral anticancer treatment) for example : fever over 38.5°C, nosebleeds and /or bleeding gums, breathlessness, respiratory difficulties, chest pain, swelling, pain or redness in the legs, digestive difficulties, insomnia, fatigue, tingling, numb fingers or toes.

D. For both groups in the study, evaluate the adherence to treatment (adherence rate in percentages).

E. Evaluate the rate of discrepancies per item : treatment started in due time, right molecule taken at the right moment, respect of days when no medication is to be taken, day when treatment is to be stopped.

ELIGIBILITY:
Inclusion Criteria:

* All patients being treated for multiple myeloma receiving their first oral anticancer treatment.
* All patients being treated for multiple myeloma by autologous peripheral stem cell graft following the Revlimid - Velcade - Dexamethazone protocol
* All patients who cannot be treated for multiple myeloma by autologous peripheral stem cell graft and who are following the Revlimid - Dexamethazone protocol
* All patients who have given written informed consent.
* All patients who have signed the consent form.
* All patients covered by a health insurance scheme

Exclusion Criteria:

* All patients requiring help at home from a nurse for taking their oral treatment
* All patients participating in another category 1 research project.
* All patients in an exclusion period determined by another study.
* All patients for whom it is impossible to give enlightened information.
* All patients who are pregnant or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Observance of treatment by patients following Revlimid - Velcade - Dexamethasone protocol who had the benefit of a Guided Clinical Pharmacy Consultation | End of treatment. Day 21 +/- 5 days
  The rate of discrepancies between the actual prescription and what the patient has noted on the daily report will be measured as a percentage.
Observance of treatment by patients following Revlimid - Dexamethazone protocol who had the benefit of the Guided Clinical Pharmacy Consultation | End of treatment. Day 28 +/- 5 days
  The rate of discrepancies between the actual prescription and what the patient has noted on the daily report will be measured as a percentage.
Observance of treatment by patients following Revlimid - Velcade - Dexamethasone protocol who did not not have the benefit of a Guided Clinical Pharmacy Consultation | End of treatment. Day 21 +/- 5 days
  The rate of discrepancies between the actual prescription and what the patient has noted on the daily report will be measured as a percentage.
Observance of treatment by patients following Revlimid - Dexamethazone protocol who did not have the benefit of the Guided Clinical Pharmacy Consultation | End of treatment. Day 28 +/- 5 days
  The rate of discrepancies between the actual prescription and what the patient has noted on the daily report will be measured as a percentage

SECONDARY OUTCOMES:
Results of the self-questionnaire for patients following the Revlimid - Velcade - Dexamethasone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  Percentage of right answers to the self-questionnaire testing patient's knowledge and understanding of treatment as explained in the guide given at the time of the consultation for patients benefitting from the guided clinical pharmacy consultation
Results of the self-questionnaire for patients following the Revlimid - Velcade - Dexamethasone protocol who did not have the benefit of the guided clinical pharmacy consultation | End of treatment. Day 21 +/- 5 days
  Percentage of right answers to the self-questionnaire testing patient's knowledge and understanding of treatment.
Results of the self-questionnaire for patients following the Revlimid - Dexamethazone protocol who benefitted from the guided clinical pharmacy consultation | End of treatment. Day 28 +/- 5 days
  Percentage of right answers to the self-questionnaire testing patient's knowledge and understanding of treatment as explained in the guide given at the time of the consultation for patients benefitting from the guided clinical pharmacy consultation
Results of the self-questionnaire for patients following the Revlimid - Dexamethazone protocol who did not have the benefit of the guided clinical pharmacy consultation | End of treatment. Day 28 +/- 5 days
  Percentage of right answers to the self-questionnaire testing patient's knowledge and understanding of treatment.
System Usability Score for patients following Revlimid - Velcade - Dexamethasone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  The System Usability Score is a set of 10 questions with a 5-point Lickert scale ranging from "I disagree" to "I completely agree". The satisfaction score ranges from 0 to 100.
System Usability Score for patients following Revlimid - Velcade - Dexamethasone protocol who did not have the benefit of the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  The System Usability Score is a set of 10 questions with a 5-point Lickert scale ranging from "I disagree" to "I completely agree". The satisfaction score ranges from 0 to 100.
System Usability Score for patients following Revlimid - Dexamethazone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 28 +/- 5 days
  The System Usability Score is a set of 10 questions with a 5-point Lickert scale ranging from "I disagree" to "I completely agree". The satisfaction score ranges from 0 to 100.
System Usability Score for patients following Revlimid - Dexamethazone protocol who did not have the benefit of the guided clinical pharmacy consultation. | End of treatment. Day 28 +/- 5 days
  The System Usability Score is a set of 10 questions with a 5-point Lickert scale ranging from "I disagree" to "I completely agree". The satisfaction score ranges from 0 to 100.
Semi-directive interview for patients following Revlimid - Velcade - Dexamethasone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  The following events are that may have affected treatment observance are noted:
  fever over 38.5°, Nosebleeds or bleeding gums, Breathlessness, respiratory difficulties, Chest pain, Swelling, pain or redness in the legs, Digestive difficulties, Insomnia, Fatigue, Tingling, Numb fingers or toes
Semi-directive interview for patients following Revlimid - Velcade - Dexamethasone protocol who did not have the benefit of the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  The following events are that may have affected treatment observance are noted:
  fever over 38.5°, Nosebleeds or bleeding gums, Breathlessness, respiratory difficulties, Chest pain, Swelling, pain or redness in the legs, Digestive difficulties, Insomnia, Fatigue, Tingling, Numb fingers or toes
Semi-directive interview for patients following Revlimid - Dexamethazone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 28 +/- 5 days
  The following events are that may have affected treatment observance are noted:
  fever over 38.5°, Nosebleeds or bleeding gums, Breathlessness, respiratory difficulties, Chest pain, Swelling, pain or redness in the legs, Digestive difficulties, Insomnia, Fatigue, Tingling, Numb fingers or toes
Semi-directive interview for patients following Revlimid - Dexamethazone protocol who did not have the benefit of the guided clinical pharmacy consultation. | End of treatment. Day 28 +/- 5 days
  The following events are that may have affected treatment observance are noted:
  fever over 38.5°, Nosebleeds or bleeding gums, Breathlessness, respiratory difficulties, Chest pain, Swelling, pain or redness in the legs, Digestive difficulties, Insomnia, Fatigue, Tingling, Numb fingers or toes
Pill-count for patients following Revlimid - Velcade - Dexamethasone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  Treatment observance rate as a percentage deduced from the number of pills prescribed and the number of pills taken.
Pill-count for patients following Revlimid - Velcade - Dexamethasone protocol who did not benefit from the guided clinical pharmacy consultation. | End of treatment. Day 21 +/- 5 days
  Treatment observance rate as a percentage deduced from the number of pills prescribed and the number of pills taken.
Pill-count for patients following Revlimid - Dexamethazone protocol who benefitted from the guided clinical pharmacy consultation. | End of treatment. Day 28 +/- 5 days
  Treatment observance rate as a percentage deduced from the number of pills prescribed and the number of pills taken.
Pill-count for patients following Revlimid - Dexamethazone protocol who did not benefit from the guided clinical pharmacy consultation. | End of treatment. Day 28 +/- 5 days
  Treatment observance rate as a percentage deduced from the number of pills prescribed and the number of pills taken.
Rate of discrepancies per item in patients on Revlimid - Velcade - Dexamethasone protocol who benefitted from the Guided Clinical Pharmacy Consultation | End of treatment. Day 21 +/- 5 days
  The following items recorded on the patient's journal - treatment begun in due time, right molecule taken at the right time, respect for days without medication, day when treatment was stopped - will be converted into a percentage rate of discrepancies.
Rate of discrepancies per item in patients on Revlimid - Velcade - Dexamethasone protocol who did not benefit from the Guided Clinical Pharmacy Consultation | End of treatment. Day 21 +/- 5 days
  The following items recorded on the patient's journal - treatment begun in due time, right molecule taken at the right time, respect for days without medication, day when treatment was stopped - will be converted into a percentage rate of discrepancies.
Rate of discrepancies per item in patients on Revlimid - Dexamethazone protocol who benefitted from the Guided Clinical Pharmacy Consultation | End of treatment. Day 28 +/- 5 days
  The following items recorded on the patient's journal - treatment begun in due time, right molecule taken at the right time, respect for days without medication, day when treatment was stopped - will be converted into a percentage rate of discrepancies.
Rate of discrepancies per item in patients on Revlimid - Dexamethazone protocol who did not benefit from the Guided Clinical Pharmacy Consultation | End of treatment. Day 28 +/- 5 days
  The following items recorded on the patient's journal - treatment begun in due time, right molecule taken at the right time, respect for days without medication, day when treatment was stopped - will be converted into a percentage rate of discrepancies.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Nîmes University Hospital, Nîmes, Occitanie
  - Dijon University Hospital Pharmacy, Dijon
  - Perpignan Hospital Center, Perpignan

IPD SHARING:
Plan to Share IPD: No